CLINICAL TRIAL: NCT05766709
Title: Investigation of Pharmacokinetics Following Administration of NNC0194-0499 and Semaglutide as Co-formulation Versus Separate Injections in Healthy Participants
Brief Title: A Research Study Comparing Blood Levels of Medicines NNC0194-0499 and Semaglutide Administered as a Combination Formulation Versus Two Separate Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NN9500-4932; U1111-1285-5065 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-02-23; First posted 2023-03-13 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Non-alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1 (Experimental): Participants will receive separate injections of NNC0194-0499 B and Semaglutide B for 24 weeks. Dose escalation manner every 4 weeks for 20 weeks (30 mg NNC0194-0499 B and 0.24 mg Semaglutide B for Weeks 1-4, 30 mg NNC0194-0499 B and 0.5 mg Semaglutide B for Weeks 5-8, 30 mg NNC0194-0499 B and 1.0 mg Semaglutide B for Weeks 9-12, 30 mg NNC0194-0499 B and 1.7 mg Semaglutide B for Weeks 13-16 and 30 mg NNC0194-0499 B and 2.4 mg Semaglutide B for Weeks 17-20). Participants will receive NNC0194-0499/Semaglutide A 40/3.20 mg/mL co-formulation at the target dose of 30/2.4 mg during the weeks 21-24 (maintenance dosing period).
  Interventions: Drug: NNC0194-0499; Drug: Semaglutide; Drug: NNC0194-0499/Semaglutide A (40/3.20 mg/mL)
- Group 2 (Experimental): Participants will receive NNC0194-0499/Semaglutide A 40/3.20 mg/mL co-formulation for 24 weeks. Dose escalation manner every 4 weeks for 20 weeks (3.1mg/0.25mg for Weeks 1-4, 6.3mg/0.5mg for Weeks 5-8, 12.5mg/1.0mg for Weeks 9-12, 21.3mg/1.7mg for Weeks 13-16 and 30mg/2.4mg for weeks 17-20). Participants will receive NNC0194-0499/Semaglutide 40/3.20 mg/mL co-formulation at the target dose of 30mg/2.4mg during the weeks 21-24 (maintenance dosing period).
  Interventions: Drug: NNC0194-0499/Semaglutide A (40/3.20 mg/mL)
- Group 3 (Experimental): Participants will receive 4 weekly injections of NNC0194-0499/Semaglutide A 40/0.33 mg/mL co-formulation at the dose level of 30mg/0.25 mg.
  Interventions: Drug: NNC0194-0499/Semaglutide A (40/0.33mg/mL)

INTERVENTIONS:
Drug: NNC0194-0499 — NNC0194-0499 will be administered subcutaneously once weekly.
  Arms: Group 1
Drug: Semaglutide — Semaglutide will be administered subcutaneously once weekly.
  Arms: Group 1
Drug: NNC0194-0499/Semaglutide A (40/3.20 mg/mL) — NNC0194-0499/Semaglutide A (40/3.20 mg/mL) co-formulation product will be administered subcutaneously once weekly.
  Arms: Group 1; Group 2
Drug: NNC0194-0499/Semaglutide A (40/0.33mg/mL) — NNC0194-0499/Semaglutide A (40/0.33mg/mL) will be administered subcutaneously once weekly.
  Arms: Group 3

SUMMARY:
Novo Nordisk is developing a combination of 2 medicines (NNC0194-0499 and semaglutide) for the treatment of nonalcoholic steatohepatitis (NASH). NASH is a serious disease where fat, inflammation and scar tissue builds up in the liver. NNC0194-0499 is a new medicine which works in the liver. Semaglutide is a well-known medicine, which is already used to treat type 2 diabetes and obesity. The study is being done to see how 2 medicines (NNC0194-0499 and semaglutide) are absorbed, transported, and eliminated from the body in a combination formulation. Participants will either get NNC0194-0499 and semaglutide in a combination formulation or the separate formulations. Which treatment participants get is decided by chance. The study will last for either 13 or 33 weeks. The duration is decided by chance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18-55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between greater than or equal to 25 and less than or equal to 35 kilogram per meter square (kg/m^2) (both inclusive)
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive method
* Participation (that is, signed informed consent) in any other interventional clinical study within 90 days before first trial product administration (Visit 2, Day 1)
* Use of prescription medicinal products or non-prescription drugs, except routine vitamins, topical medication, highly effective contraceptives and occasional use of paracetamol, acetylsalicylic acid within 14 days before first trial product administration (Visit 2, Day 1)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
AUC 0-168 hour (h), 0499, steady state (SS): Area under the NNC0194-0499 concentration time curve during a dosing interval (0-168 hours) at steady state after dosing of NNC0194-0499 in combination with semaglutide | Day 134 (pre-dose) to Day 141 (168 hours post-dose)
  Measured as nanomoles*hours per liter (nmol*h/L)
AUC 0-168h,sema,SS: Area under the semaglutide concentration time curve during a dosing interval (0-168 hours) at steady state after dosing of NNC0194-0499 in combination with semaglutide | Day 134 (pre-dose) to Day 141 (168 hours post-dose)
  Measured as nmol*h/L
Cmax, 0499, SS: Maximum concentration of NNC0194-0499 at steady state after dosing of NNC0194-0499 in combination with semaglutide | Day 134 (pre-dose) to Day 141 (168 hours post-dose)
  Measured as nanomoles per liter (nmol/L)
Cmax,sema, SS: Maximum concentration of semaglutide at steady state after dosing of NNC0194-0499 in combination with semaglutide | Day 134 (pre-dose) to Day 141 (168 hours post-dose)
  Measured as nmol/L

SECONDARY OUTCOMES:
AUC 0-168h, 0499, SS: Area under the NNC0194-0499 concentration-time curve during a dosing interval (0-168 hours) at steady state after dosing of NNC0194-0499 in combination with semaglutide | Day 22 (pre-dose) to Day 29 (168 hours post-dose)
  Measured as nmol*h/L
AUC 0-168h, sema , SS: Area under the semaglutide concentration-time curve during a dosing interval (0-168 hours) at steady state after dosing of semaglutide in combination with NNC0194-0499 | Day 22 (pre-dose) to Day 29 (168 hours post-dose)
  Measured as nmol*h/L
Cmax, 0499, SS: Maximum concentration of NNC0194-0499 at steady state after dosing of NNC0194-0499 in combination with semaglutide | Day 22 (pre-dose) to Day 29 (168 hours post-dose)
  Measured as nmol/L
Cmax, sema , SS: Maximum concentration of semaglutide at steady state after dosing of semaglutide in combination with NNC0194-0499 | Day 22 (pre-dose) to Day 29 (168 hours post-dose)
  Measured as nmol/L
Number of treatment emergent adverse events | Day 1 (post-dose) to Day 197 (Groups 1 and 2) and Day 1 (post-dose) to Day 57 (Group 3)
  Measured as count of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept.2834, Study Director — Novo Nordisk A/S
Locations (1):
- Altasciences Company Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com